CLINICAL TRIAL: NCT03996499
Title: Myocardial Perfusion, Coronary Flow Reserve and Kinetic Analysis During Dobutamine Stress Echocardiography
Acronym: TRIPLESTRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TRIPLESTRESS
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Echocardiography, Stress

STUDY DESIGN:
Intervention Model Description: The course of the examination corresponds to the welcome of the patient, the search for contraindications and the performance of the stress ultrasound. During this stress ultrasound, the 3 indices (segmental kinetics, coronary reserve and myocardial perfusion) will be analyzed. The duration of the ultrasound is not lengthened (examination time: 20 minutes).
  The evaluation of the myocardial perfusion is carried out thanks to the use of the "flash", modality not being part of the usual care.
  Indeed, during the examination, the power of the probe will be increased to evaluate the myocardial perfusion. The bubbles of the contrast medium are destroyed by applying a "flash", that is to say a transient increase in the power of the ultrasonic beam. Systole after systole, on a recorded loop, the filling rate of the myocardium, which depends on the myocardial blood flow, is analyzed. The evaluation of the infusion is visual and qualitative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress echocardiography (Experimental): The course of the examination corresponds to the welcome of the patient, the search for contraindications and the performance of the stress ultrasound. During this stress ultrasound, the 3 indices (segmental kinetics, coronary reserve and myocardial perfusion) will be analyzed. The duration of the ultrasound is not lengthened (examination time: 20 minutes).
  The evaluation of the myocardial perfusion is carried out thanks to the use of the "flash", modality not being part of the usual care.
  Indeed, during the examination, the power of the probe will be increased to evaluate the myocardial perfusion. The bubbles of the contrast medium are destroyed by applying a "flash", that is to say a transient increase in the power of the ultrasonic beam. Systole after systole, on a recorded loop, the filling rate of the myocardium, which depends on the myocardial blood flow, is analyzed. The evaluation of the infusion is visual and qualitative.
  Interventions: Diagnostic Test: Stress echocardiography

INTERVENTIONS:
Diagnostic Test: Stress echocardiography — The course of the examination corresponds to the welcome of the patient, the search for contraindications and the performance of the stress ultrasound. During this stress ultrasound, the 3 indices (segmental kinetics, coronary reserve and myocardial perfusion) will be analyzed. The duration of the ultrasound is not lengthened (examination time: 20 minutes).
  The evaluation of the myocardial perfusion is carried out thanks to the use of the "flash", modality not being part of the usual care.
  Indeed, during the examination, the power of the probe will be increased to evaluate the myocardial perfusion. The bubbles of the contrast medium are destroyed by applying a "flash", that is to say a transient increase in the power of the ultrasonic beam. Systole after systole, on a recorded loop, the filling rate of the myocardium, which depends on the myocardial blood flow, is analyzed. The evaluation of the infusion is visual and qualitative.

SUMMARY:
Stress echocardiography is a screening test for coronary heart disease that already has good sensitivity and specificity (both around 70%). This examination is mainly offered to stable patients, consulting externally, in order to detect ischemic heart disease in the same way as would a myocardial scintigraphy or MRI stress. This examination is an echocardiographic modality consisting in visualizing and analyzing the modifications of the contraction of the cardiac muscle during a stress constituted by an effort or by injection of certain drugs. Stress echocardiography is performed by injection of drugs to reproduce the conditions of the effort. The products used to perform this examination are initially an intravenous infusion of dobutamine, atropine whose effect is to increase the heart rate, and in a second time, an intravenous infusion of beta-blockers or a bradycardic calcium channel blocker at the end of the procedure whose effect is to slow down the heart rate.

The use of echographic contrast medium, allowing a better visibility, is recommended for the realization of a stress ultrasound, since the echogenicity is judged insufficient on two segments (segmentation of the left ventricle in 17 segments).

The analysis of dobutamine stress echocardiography currently relies solely on the analysis of segmental kinetics, namely the quality of the thickening of the endocardium. When segmental kinetics are abnormal, patients benefit from a coronary CT scan or coronary angiography to visualize all the coronary arteries and to check whether there is a narrowing of the arteries.

Moreover, stress echocardiography performed using a contrast medium makes it possible to analyze two other indices in addition to segmental kinetics.

Thus, the second parameter that can be analyzed corresponds to the Coronary Flow Reserve measurement, thanks to the easy identification of the Doppler flow in the anterior interventricular at rest and peak of dobutamine. The coronal reserve is well validated with adenosine, but much less well known under dobutamine.

The third parameter that can be analyzed is myocardial perfusion. By using appropriate settings, it is possible to see the microbubbles in the thickness of the myocardium. These bubbles are then destroyed by an ultrasonic flash of high mechanical index. This results in the destruction of all intra-myocardial bubbles. The analysis of the myocardial perfusion is based on the rate of reappearance of these bubbles (through the coronary arteries) at rest and peak stress. In case of significant stenosis or coronary occlusion, there is a delay or complete absence of perfusion in the territory concerned.

Joint analysis of segmental kinetics, coronary reserve and myocardial perfusion has already been described with adenosine, but not with dobutamine. Studies in the literature suggest that the analysis of coronary reserve on the one hand, and myocardial perfusion on the other hand would increase the sensitivity and specificity of the examination. In addition, other studies suggest that among the tests considered normal for segmental kinetics analysis, there are patients with myocardial perfusion abnormality and / or coronary reserve abnormality that strike (s) on prognosis (alteration of the coronary microcirculation).

This is why it seems interesting to compare the results of these 3 indices obtained during stress echocardiography under dobutamine.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient referred for stress echography in the context of a cardiovascular assessment or for suspicion of coronary disease
* Patient whose echogenicity requires the use of an ultrasound contrast product (SONOVUE®) according to European Society of Cardiology recommendations
* Patient affiliated with a health insurance plan
* Francophone patient
* Patient able to give free, informed and written oral consent

Exclusion Criteria:

* People in emergency situations (recent acute coronary syndromes) who can not express their prior consent
* Patient with an allergy to any of the products used
* Patient for whom it is impossible to obtain a theoretical maximum frequency (continued beta-blocker treatment, chronotropic insufficiency)
* Pregnant woman
* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the combined analysis | Day 1
  This is to measure the sensitivity of segmental kinetics, coronary reserve and myocardial perfusion compared to simple segmental kinetic analysis alone to detect coronary artery disease.
Specificity of the combined analysis | Day 1
  This is to measure the specificity of segmental kinetics, coronary reserve and myocardial perfusion compared to simple segmental kinetic analysis alone to detect coronary artery disease.

SECONDARY OUTCOMES:
Rate of complications | Year 2
  This is to measure rate of cardiovascular mortality, hospitalization for acute coronary syndromes or emergency coronary revascularization in patients with negative examination on 1, 2 or 3 index.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe P GARCON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France